CLINICAL TRIAL: NCT02321852
Title: Randomized Placebo Controlled Phase II Cross Over Study on the Influence of Triflusal on Cognitive Functions in Healthy Participants
Brief Title: Influence of Triflusal on Cognitive Functions in Healthy Subjects
Acronym: Tribunal-Basel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014DR2154
Record Dates: First submitted 2014-12-02; First posted 2014-12-22 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — triflusal; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum/Placebo (Experimental): This group will start with triflusal and after washout will receive placebo
  Interventions: Drug: Triflusal; Drug: Placebo
- Placebo/Verum (Experimental): This group will start with placebo and will receive triflusal after washout.
  Interventions: Drug: Triflusal; Drug: Placebo

INTERVENTIONS:
Drug: Triflusal — Once daily oral administration of 600 mg triflusal Disgren® for 7 days.
  Other Names: Disgren®
Drug: Placebo — Once daily oral administration of placebo mannitol for 7 days
  Other Names: Mannitol

SUMMARY:
The purpose of this study is to investigate the effects of the eNOS activating agent triflusal on episodic memory and cognitive functions in healthy participants.

DETAILED DESCRIPTION:
Randomised, placebo controlled, double blind, cross-over design

Primary study outcomes are:

Performance in picturial and verbal memory tasks.

Main secondary outcomes are: Performance in working memory and cognitive tasks and influence on mood, depression and anxiety and motivation.

Once daily oral administration of placebo mannitol for 7 days in a cross-over trial with a washout period of at least 14 days between the two periods. Each participant will take triflusal as well as placebo

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male or female
* Normotensive
* BMI between 20 and 27 kg/m2
* Aged between 18 and 40 years
* Native or fluent German-speaking
* Caucasian
* Female practicing safe contraception

Exclusion Criteria:

* Acute or chronic psychiatric or somatic disorder
* Any contraindication against aspirin or other NSAIDS
* History of coagulation disease
* History of gastrointestinal disease
* Laboratory exclusion criteria: values of blood count, blood chemistry and coagulation status outside normal range
* Pathological ECG
* Pregnancy, breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in performance in episodic memory task as assessed by a picturial memory task between placebo and verum at two different timepoints | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Picture task as described in (de Quervain, Kolassa et al. 2007). Number of correctly remembered pictures is counted.
Change in performance in episodic memory task as assessed by a verbal memory task between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Verbal task as described in ( de Quervain, Henke et al. 2003). Number of correctly remembered words is counted.

SECONDARY OUTCOMES:
Change in performance in working memory task between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Working memory as assessed by digit span task. Number of correctly remembered digitsis counted.
Change in performance in a cognitive task between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Cognitive performance as assessed by BOMAT matrix reasoning task. Number of correct solutions is counted.
Mood state changes between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Mood state as assessed by self-rating instrument MDBF. Total score is calculated by summing the answers of nine items.
Changes in depressive symptoms between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Depressive symptoms as assessed by self-rating instrument MADRS.Total score is calculated by summing the answers of nine items.
Change in anxiety symptoms between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Anxiety symptoms as assessed by self-rating instrument STAI-G from X1 (state). Total score is calculated by summing the answers.
Change in motivation between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 2: 24 h after last medication.
  Motivation is assessed by a visual analogue scale ranging between 0 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique De Quervain, MD, Principal Investigator — Division of Cognitive Neuroscience University of Basel
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Basel, Switzerland